CLINICAL TRIAL: NCT02552524
Title: Study of the Effect of an Active rTMS Session in Pathological Gamblers: Impact on Craving and Severity of These Behaviors
Brief Title: Effect of rTMS in Pathological Gamblers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1201091; 2012-A01013-40 (Other: ANSM)
Record Dates: First submitted 2015-09-11; First posted 2015-09-17 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Pathological Gambler
Keywords: pathological gambling; rTMS; cognitive tests; autonomic nervous system; craving
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rTMS active then rTMS placebo (Experimental): A 20 minute session of rTMS active at the frequency of 10 Hz then, 7 days later, a 20 minute session of rTMS placebo (rTMS active then rTMS placebo).
  Patient will also have cognitive tests before and after rTMS session and HRV recording during visit.
  Interventions: Device: rTMS active then rTMS placebo
- rTMS placebo then rTMS active (Experimental): A 20 minute session of rTMS placebo then, 7 days later, a 20 minute session of rTMS active at the frequency of 10 Hz (rTMS placebo then rTMS active).
  Patient will also have cognitive tests before and after rTMS session and HRV recording during visit
  Interventions: Device: rTMS placebo then rTMS active

INTERVENTIONS:
Device: rTMS active then rTMS placebo — A 20 minute session of rTMS active at the frequency of 10 Hz then, 7 days later, a 20 minute session of rTMS placebo
  Arms: rTMS active then rTMS placebo
Device: rTMS placebo then rTMS active — A 20 minute session of rTMS placebo then, 7 days later, a 20 minute session of rTMS at the frequency of 10 Hz
  Arms: rTMS placebo then rTMS active

SUMMARY:
The gambling problem is characterized by a loss of control and an excessive focus on the gambling practice. Currently, the treatment of pathological gamblers is often complex and multidimensional, it notably includes psychological techniques including cognitive behavioral therapy and the use of psychotropic drugs.

In pathological gambling and addictions, craving (or urge to play) and loss of control are two essential clinical elements. The neurobiological level, they are associated with a dysfunction of dorsolateral prefrontal cortex (DLPFC) (Goldstein et al, 2001, Volkow and Goldstein, 2002).

One therapeutic avenues explored in addictions is repeated transcranial magnetic stimulation (rTMS).

DETAILED DESCRIPTION:
Patients included in this study will have:

* An anatomical brain MRI (30 minutes).
* Two 20 minute sessions of rTMS (placebo and active) of the left DLPFC, at the frequency of 10 Hz.
* Visual Analogue Scale measuring their desire to gamble before and after a gambling video and test measuring their gambling behavior during the last 7 days (PG-YBOCS).
* Cognitive tests, to be carried out on a computer before and immediately after rTMS sessions.
* Recording heart rate variability (HRV) to measure the autonomic nervous system (ANS) activity

As it is a pilot study, the investigators don't have sufficient data to calculate statistical power and number of participants. The investigators based on previous studies evaluating one rTMS session on craving in SUD and used a crossover design to generate greater power.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of pathological gambling (DSM IV criteria)
* First-time consultants.
* Without psychotropic treatment or treatment with a stable and unchanged for over a month.

Exclusion Criteria:

* Presence of ferromagnetic material or devices implanted neurostimulation in close contact with the coil
* Pregnant women and patients with hearing disorders
* Personal history of epilepsy (untreated or poorly balanced)
* Focal brain injury, whatever its origin (vascular, traumatic, tumor or infectious)
* History of head trauma with loss of consciousness,
* Administration of drugs or substances lowering the seizure threshold
* Sleep deprivation, jet lag, or drug withdrawal.
* Participants with a problem of uncorrected visual acuity.
* Other current addiction (except tobacco, for reasons of feasibility).
* Current Psychiatric comorbidity
* Treatment psychotropic introduced or changed for less than a month.
* Subjects with atrial fibrillation, with a pacemaker and / or receiving antiarrhythmic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Assessing cue-induced craving | After the session of rTMS (Day 2)
  Scores on visual analog scales assessing craving just after a gambling video

SECONDARY OUTCOMES:
Game behavior | Day 2
  Scores at the PG-YBOCS (obsessions-compulsions scale Yale-Brown (Y-BOCS), adapted for pathological gambling) (PG-YBOCS) (Pallanti et al., 2005)) assessing the severity of gambling behavior over the past week
Cognitive tests | Day 2
  Reaction time and number of errors at Go-Nogo, Flexibility task and Iowa Gambling test
ANS activity | Day 2
  Indice HF, LF and LF/HF, heart rate; during gambling video

CONTACTS AND LOCATIONS:
Overall Officials: Aurelia GAY, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gay A, Boutet C, Sigaud T, Kamgoue A, Sevos J, Brunelin J, Massoubre C. A single session of repetitive transcranial magnetic stimulation of the prefrontal cortex reduces cue-induced craving in patients with gambling disorder. Eur Psychiatry. 2017 Mar;41:68-74. doi: 10.1016/j.eurpsy.2016.11.001. Epub 2017 Feb 3. PMID 28049084